CLINICAL TRIAL: NCT00870233
Title: Electronic Patient-Reported Outcomes From Home in Patients Recovering From Major Gynecologic Cancer Surgery: Measuring Symptoms and Health-related Quality of Life
Brief Title: Outcomes From Home in Patients Recovering From Major Gynecologic Cancer Surgery: Measuring Symptoms and Health-related Quality of Life
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-155
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-07

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cancer; Uterine Cancer; Vaginal Cancer; Vulvar Cancer
Keywords: Gynecologic cancers; Quality of Life; 08-155; Surgery
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- GYN pts undergoing surgery: This study will assess patient use of WEBCORE, an online system designed for cancer patients to self-record toxicity-related symptoms based on NCI Common Terminology Criteria for Adverse Events and global quality of life (QoL) by European Organization for Research and Treatment of Cancer (EORTC QLQ-C30).
  Interventions: Behavioral: online platform WEBCORE

INTERVENTIONS:
Behavioral: online platform WEBCORE — Enrollees will be sent weekly email reminders to login to WEBCORE from home. Participants will be expected to complete the questionnaire once pre-operatively and then weekly starting 7 days after surgery until the 6-week post-operative period has ended.
  Other Names: If an enrolled patient fails to login and self-report within 24 hours of; the automated reminder, a second reminder email will be sent. If the; patient again fails to respond, a backup telephone call to the patient; will be made by the clinical research fellow coordinating this study.; The back-up phone call will be made within a week of the initial missed; questionnaire. If the patient is unreachable, a total of 3 attempts will; be made to reach the patient.

SUMMARY:
This study is being done to see if most patients are willing and able to report how they are feeling after surgery using the internet, and if this information can help doctors and nurses detect concerning symptoms after surgery.

This study uses a special new website called WEBCORE. Patients can logon to WEBCORE and answer questions about how they are feeling. Then, doctors and nurses can look at this information during clinic appointments. We are doing this study to see if WEBCORE is a helpful way for us to keep track of information about how patients are feeling and quality of life. If WEBCORE is helpful, we will use it in the future to collect more information about patients' symptoms and quality of life. We can use what we learn to help find better ways of helping patients to prepare for what they will go through while they recover from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older
* Participants must be able to provide informed consent
* Participants must be scheduled to undergo laparotomy for presumed or known gynecologic cancer
* The assessments were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the tests. Participants must be able to speak and read English fluently
* Participants must have access to a home computer, have a personal email account, and check email at least once weekly by self-report

Exclusion Criteria:

* Patients who have a cognitive or psychiatric deficit resulting in an inability to provide meaningful informed consent, as judged by the consenting professional, and/or as noted in the medical record
* Patients who are undergoing pelvic exenterative surgery (with the exception of patients undergoing modified pelvic exenteration in the context of debulking for ovarian or uterine cancer).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparotomy for presumed or confirmed gynecologic malignancy at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-03-24 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GYN Pts Undergoing Surgery
Started | 120
Completed | 96
Not Completed | 24
Not completed — Withdrawal by Subject | 18
Not completed — Did not undergo laparotomy | 3
Not completed — Incompatible internet browser | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | GYN Pts Undergoing Surgery
Number analyzed (Participants) | 120
Age, Continuous [Median (Full Range); unit: years] | 55 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 113
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 105
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Electronic Capture of Patient-reported Symptoms From Home Following Major Gynecologic Cancer Surgery
Time Frame: once pre-operatively and then weekly starting 7 days after surgery until the 6-week post-operative period has ended.
Measure: Count of Participants; unit: Participants
Arm/Group | GYN Pts Undergoing Surgery
Number analyzed (Participants) | 120
Participants
  Requested to be removed from study | 18
  Did not undergo lapartomy | 3
  Incompatible internet browser | 2
  Died | 1
  Completed preoperative session in STAR | 69
  Didn't complete preop, completed other surveys | 27

2. Secondary Outcome: Feasibility of Online Symptom Self-reporting in the Early Postoperative Period, and Clinician Perceptions of Its Potential Value in Routine Outpatient Post-operative Cancer Care.
Time Frame: once pre-operatively and then weekly starting 7 days after surgery until the 6-week post-operative period has ended
Population: Nurses who participated in the study
Measure: Count of Participants; unit: Participants
Groups:
- Study Nurse Clinicians: Email alerts were sent to study nurses when concerning participant responses were entered. The nurse assessments of STAR's usefulness were measured via an exit survey. Alerts were considered concerning according to pre-specified limits set by the Gynecologic Oncology Service. This is the same system presently used to triage patient phone calls. Any actions taken by the nurses in response to these alerts were recorded. However, specific responses were not required. Patients were encouraged to call their physician's office if medical attention was needed, as there was no regularly scheduled monitoring of information entered into the STAR system.
Arm/Group | Study Nurse Clinicians
Number analyzed (Participants) | 9
Participants
  Left MSK before close of study | 3
  Did not complete Clinician Exit Survey | 2
  Reported increased workload bc of STAR system | 4

3. Secondary Outcome: To Evaluate the Impact of Online Symptom Self-reporting on Patient Care Processes as Measured by the Number of Telephone Calls Between Nurses and Patients,Resulting Interventions and Patient Satisfaction With Care Delivery.
Time Frame: two years
Population: Data were not collected
Arm/Group | GYN Pts Undergoing Surgery
Number analyzed (Participants) | 0

4. Secondary Outcome: Most Commonly Reported and Most Distressing Symptoms Reported by Patients After Gynecologic Cancer Surgery Using the STAR System
Description: The percentage of symptoms generated by patients on protocol
Time Frame: weekly starting 7 days after surgery until the 6-week post-operative period
Measure: Number; unit: percentage of symptoms
Arm/Group | GYN Pts Undergoing Surgery
Number analyzed (Participants) | 120
percentage of symptoms
  ECOG Performance Status | 15
  Nausea | 14
  Fatigue | 12
  Trouble with Strenuos Activities | 17
  Constipation | 11
  Pain | 11

ADVERSE EVENTS:
Time Frame: Up to 16 weeks (between 6-8 weeks post surgery)
Arm/Group | GYN Pts Undergoing Surgery
All-Cause Mortality (participants affected / at risk) | 27/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 85/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GYN Pts Undergoing Surgery (N=120)
ECOG Performance Status (General disorders) | 17
Nausea (Gastrointestinal disorders) | 16
Fatigue (General disorders) | 13
Pain (General disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Wound complication (Injury, poisoning and procedural complications) | 7
Fever (General disorders) | 6
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT00870233/Prot_SAP_000.pdf